CLINICAL TRIAL: NCT00543595
Title: MK0916 in Patients With Type 2 Diabetes and Metabolic Syndrome (0916-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0916-005; 2007_643
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — MK-0916

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0916

SUMMARY:
This study will test the safety and effectiveness of MK0916 in patients with Type 2 Diabetes Mellitus and Metabolic Syndrome.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes
* 18 to 65 years of age

Exclusion Criteria:

* History of Type 1 Diabetes Mellitus
* Have been treated with insulin in the past 8 weeks
* On a weight loss program and have ongoing weight loss
* Taking weight loss medication
* Have had surgery requiring general anesthesia in the past 30 days or have a planned surgery
* Have taken another investigational drug in the last 8 weeks
* Have active liver disease
* Have a history of major surgery involving gastric or intestinal bypass

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Feig PU, Shah S, Hermanowski-Vosatka A, Plotkin D, Springer MS, Donahue S, Thach C, Klein EJ, Lai E, Kaufman KD. Effects of an 11beta-hydroxysteroid dehydrogenase type 1 inhibitor, MK-0916, in patients with type 2 diabetes mellitus and metabolic syndrome. Diabetes Obes Metab. 2011 Jun;13(6):498-504. doi: 10.1111/j.1463-1326.2011.01375.x. PMID 21272190